CLINICAL TRIAL: NCT04304027
Title: Feasibility Evaluation of a Tailored Exercise Intervention to Manage Fatigue in Progressive Multiple Sclerosis
Brief Title: Exercise to Manage Fatigue in Progressive Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Glasgow Caledonian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19/WS/0140
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-01

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Exercise; Fatigue
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tailored exercise intervention (Experimental): 8 weeks of aerobic interval training at moderate intensity which is modified according to the levels of self-reported fatigue
  Interventions: Other: Tailored exercise intervention
- Standard exercise intervention (Active Comparator): 8 weeks of aerobic interval training at a moderate intensity
  Interventions: Other: Standard exercise intervention
- Usual care control (No Intervention): Participants in the usual care control group will continue to receive their standard care independent of this study

INTERVENTIONS:
Other: Tailored exercise intervention — 2x 30 minute aerobic interval training per week for 8 weeks - sessions involve 6 intervals cycling for 2 minutes at target heart rate reserve followed by 2 minutes working rest (target heart rate reserve may vary between sessions depending on the level of self-reported fatigue)
  Arms: Tailored exercise intervention
Other: Standard exercise intervention — 2x 30 minute aerobic interval training per week for 8 weeks - sessions involve 6 intervals cycling for 2 minutes at >70% heart rate reserve followed by 2 minutes working rest
  Arms: Standard exercise intervention

SUMMARY:
Fatigue is one of the most common and debilitating symptoms of Multiple Sclerosis (MS). Exercise is suggested as a way to improve fatigue, but it is not clear what the effects of exercise are on fatigue - especially in people with progressive MS. Therefore, this study aims to test the feasibility of a tailored exercise programme to help improve fatigue in people with progressive MS. To do this people with progressive MS who are experiencing fatigue will be randomly allocated to receive either a tailored exercise programme, a standard exercise programme, or their usual care. Both exercise programmes will be 8 weeks long and require participants to attend Falkirk Community Hospital twice a week. The standard exercise programme involves a moderate intensity interval training session using a stationary exercise bike. The tailored exercise programme is similar to the standard exercise programme, as participants will be prescribed the same type and duration of exercise; however, the difference between the 2 programmes is that the intensity of exercise performed during each session of the tailored exercise programme is dictated by the participant's level of fatigue. Participants will complete an exercise test, walking test, and questionnaires relating to fatigue, quality of life, depression and anxiety, sleep quality, and cognition before and 1 week after completing the exercise programme.

DETAILED DESCRIPTION:
This study aims to evaluate the feasibility of delivering a tailored exercise intervention to manage fatigue in people with progressive forms of MS. To do this, a randomised controlled trial design will be used to assess the feasibility of delivering a tailored exercise intervention to manage fatigue in people with progressive forms of MS in comparison to a standard (untailored) exercise group and usual care control group.

This study aims to recruit up to 45 people with progressive MS who are experiencing moderate-severe levels of fatigue from MS clinics and outpatient physiotherapy services within NHS Forth Valley. Participants will be randomly allocated to receive either the tailored exercise programme, the standard exercise programme, or their usual care. All outcome measures will be recorded at baseline and post-intervention.

Both exercise programmes will require participants to attend Falkirk Community Hospital twice a week for 8 weeks - therefore, participants will receive 16 exercise sessions in total. All exercise sessions will be supervised by a physiotherapist and they will provide participants with any support that is required. The standard exercise programme involves aerobic-based interval training delivered on a bicycle ergometer. Each exercise session will be 30 minutes in duration, and will be broken down into a 3 minute warm-up, 24 minutes of interval training, and a 3 minute cool-down. During the interval training component, participants will be asked to perform 6 intervals that require them to exercise at a moderate intensity (>70% heart rate reserve) for 2 minutes followed by 2 minutes of recovery.

The tailored exercise programme is similar to the standard exercise programme - participants will still be required to attend Falkirk Community Hospital twice a week for 8 weeks, and they will perform the same type and duration of exercise as the standard exercise programme. However in order to tailor exercise to fatigue, participants will be asked to rate their current levels of fatigue before exercising - this rating will then be compared to the baseline score. If the participant's fatigue is worse, they will be offered the option of performing a lower intensity of exercise for that specific session (>50% heart rate reserve). In addition, participants will also be asked to monitor their fatigue in a symptom diary for 2 days following each exercise session. If fatigue is worsened by exercise and remains elevated for 2 days after 2 consecutive exercise sessions, then they will also be offered the option of performing the lower intensity exercise prescription.

Participants in the usual care control group will continue to receive their standard care independent of this study. Participants will also receive an information booklet about fatigue that is freely available from the UK MS Society. This booklet provides general information about MS-related fatigue, strategies to self-monitor and self-manage symptoms, and directs them to contact health professionals involved in their care for support if required.

ELIGIBILITY:
Inclusion Criteria:

* Neurologist-confirmed diagnosis of MS and a progressive form of the disease (either secondary or primary progressive)
* Self-report of moderate-severe fatigue in the last 7 days at screening by indicating that their fatigue is six or more when answering the following "have you had fatigue in the last seven days: between 0 (no fatigue) and 10 (extremely fatigued).
* Moderate level of disability to allow for participants to use the bicycle ergometer (indicated by an Expanded Disability Status Scale score of between ≥4 and ≤6.5)
* Be willing and able to attend Falkirk Community Hospital, twice a week for 8 consecutive weeks to receive the intervention.

Exclusion Criteria:

* A neurologist confirmed relapse of MS within the past three months
* Commenced or had a change in MS disease modifying treatment within the past six months
* Unable to provide informed consent
* Concurrently participating in another intervention trial
* Diagnosed with any of the following conditions which may also cause high levels of fatigue: anaemia, inflammatory rheumatic disease, hypothyroidism, cancer
* Cardiovascular event in the past year including but not limited to: myocardial infarction, transient ischaemic attack or cerebrovascular accident
* Diagnosis of cardiovascular, respiratory, or metabolic disease that would prevent participants from safely performing exercise including but not limited to: angina, heart failure, uncontrolled hypertension, peripheral vascular disease, chronic obstructive pulmonary disease, diabetes mellitus
* Prescription of the following medication: beta blockers, vasodilators, ACE inhibitors, diuretics or any other medication that may cause exercise induced hypotension
* Significant co-morbidity such as significant musculoskeletal or neurological conditions other than MS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Intervention tolerance | Weeks 1-8
  Participants will record the severity of fatigue before and for 48-hours following each exercise session using a Numerical Rating Scale
Intervention adherence | Weeks 1-8
  Adherence will be determined by recording the proportion of exercise sessions that each participant attends, whether the participant completes the prescribed exercise duration during each session, and whether the participant is able to reach and maintain the prescribed target heart rate
Intervention acceptability | Week 8
  The participants' views of the study procedures will be explored using an online survey. The survey contains questions relating to the content of the exercise/control groups, relevance of outcome measures included, the perceived positive/negatives of the intervention, and ways to improve the study design

SECONDARY OUTCOMES:
Fatigue Severity Scale | Baseline, 8 weeks
  Self-reported questionnaire measuring the severity of fatigue
Modified Fatigue Impact Scale | Baseline, 8 weeks
  Self-reported questionnaire measuring the impact of fatigue on physical, cognitive, and psychosocial function
Aerobic capacity | Baseline, 8 weeks
  Aerobic capacity estimated using the YMCA sub-maximal bicycle ergometer test
Multiple Sclerosis Impact Scale | Baseline, 8 weeks
  Self-reported questionnaire measuring the physical and psychological impact of Multiple Sclerosis
Hospital Anxiety and Depression Scale | Baseline, 8 weeks
  Self-reported questionnaire measuring the severity of anxiety and depression
Pittsburgh Sleep Quality Index | Baseline, 8 weeks
  Self-reported questionnaire measuring sleep quality
Symbol Digits Modalities Test | Baseline, 8 weeks
  Cognitive screening tool which measures processing speed
Six Minute Walk Test | Baseline, 8 weeks
  Measurement of the maximum walking distance covered during 6 minutes
Energy Cost of Walking | Baseline, 8 weeks
  Estimation of oxygen consumption per meter walked during the six minute walk test measured using Cosmed K4 portable oxygen telemetry system

CONTACTS AND LOCATIONS:
Overall Officials: Scott Rooney, PhD, Principal Investigator — Glasgow Caledonian University
Locations (1):
- Falkirk Community Hospital, Falkirk, United Kingdom

IPD SHARING:
Plan to Share IPD: No